CLINICAL TRIAL: NCT05481892
Title: Remote Monitoring for Equity in Advancing Control of Hypertension (REACH)
Brief Title: Remote Monitoring for Equity in Advancing Control of Hypertension
Acronym: REACH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01HL159372 (NIH); R01HL159372 (NIH)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: Blood pressure; Telehealth; Telemedicine; Patient generated health data; Remote patient monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Cellular Home blood pressure (BP) monitoring with minimal support (Experimental): Patients will be instructed to write down their blood pressures (BP) in a BP log that will be provided to them at the time of enrollment. Study staff will access the patient's home BP measurements on the BP device dashboard and send a summary of the home BP measurements (mean, median, % of BP measurements at goal) to the primary care provider in a telephone encounter (TE) 3 to 5 days prior to the next scheduled visit.
  Interventions: Device: Cellular Home blood pressure (BP) monitoring
- Cellular Home blood pressure (BP) monitoring with pharmacist support for treatment intensification (Active Comparator): For patients randomized to this intervention arm, a pharmacist will review the home blood pressure (BP) measurements and use an evidence-based algorithm to make recommendations for medication intensification. If the patient has a primary care provider (PCP) appointment within 2 weeks, the pharmacist will send a telephone encounter (TE) with BP measurements and medication recommendations to the PCP 3 -5 days prior to the scheduled appointment. If the patients has no appointment scheduled within two weeks, the pharmacist will call the patient and prescribe medication intensification if the patient is amenable.
  Interventions: Device: Cellular Home blood pressure (BP) monitoring
- Non-randomized usual care (No Intervention): To compare the two intervention arms with usual care, investigators will extract electronic health record (EHR) data on active San Francisco Health Network (SFHN) adult patients (age 18+) with diagnosis of hypertension who made at least one primary care visit during the study period.

INTERVENTIONS:
Device: Cellular Home blood pressure (BP) monitoring — Patients receiving intervention will receive cellular home blood pressure (BP) monitoring devices. Some patients will also receive pharmacist support for treatment intervention.
  Arms: Cellular Home blood pressure (BP) monitoring with minimal support; Cellular Home blood pressure (BP) monitoring with pharmacist support for treatment intensification

SUMMARY:
The goal of this study is to support patients with hypertension self-management using both home blood pressure monitors and digital messaging programs. The investigators will first engage patients with technology training to use home monitors, online portal websites to view their medical record information online, and texting and mobile phone applications. Then investigators will assess the effectiveness of home blood pressure monitors and enhanced patient-clinician digital communication on blood pressure control during a 12-month intervention.

DETAILED DESCRIPTION:
This study aims to launch an effectiveness-implementation hybrid randomized trial to adapt a multi-faceted hypertension (HTN) management program shown to work in integrated healthcare delivery systems to a safety net healthcare system, San Francisco Health Network (SFHN). In Aim 1 of this study, investigators will offer patients brief in-person training to support their use of the online patient portal and basics about text messaging. Investigators will examine pre-post training changes in technology use overall as well as by specific patient subgroups with known differences in technology uptake. In Aim 2 investigators will conduct a three-arm randomized controlled trial to compare varying levels of implementation support: 1) cellular-enabled blood pressure (BP) monitors (with minimal implementation support), 2) cellular-enabled BP monitors with protocol-based implementation support (text reminders for patients; aggregated BP summaries sent to primary care providers), and 3) cellular-enabled BP monitors and pharmacist-led support (pharmacist coaching and independent medication adjustments). In Aim 3 investigators will use a mixed methods approach to evaluate key implementation outcomes, guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, of adapting an existing, evidence-based home BP monitoring program.

ELIGIBILITY:
Inclusion Criteria:

* English-and Spanish-speaking patients
* Patient within the San Francisco Health Network (SFHN)
* Has seen primary care provide within the past 2 years
* Uncontrolled hypertension (HTN) in the HTN registry
* Complete Aim 1 training, in addition to patients who have not completed Aim 1 training
* Over the age of 18

Exclusion Criteria:

* Under the age of 18
* Controlled HTN

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | 6 months
  We will use clinic-based assessment of SBP as the primary outcome of interest, using all SBP measurements during any outpatient encounter in the 6 months prior to enrollment in the study and the 6 months during the active intervention period. Blood pressure (BP) is collected routinely during all patient encounters in our system, using a standardized BP measurement protocol that requires the use of automated BP machines at primary clinics broadly implemented as part of ongoing, previously described, qualify improvement efforts.

SECONDARY OUTCOMES:
Medication intensification | 6 months
  We will review prescribing patterns for anti-hypertensive medications for each patient in the trial. This will be measured as total proportion of patients with medication intensification (new medication or increased dosage) over the study period.
Blood Pressure (BP) control | 6 months
  We will define BP control as Systolic blood pressure (SBP) <140mmg and Diastolic blood pressure (DBP) <90 mmHg in secondary analyses. This BP control analysis will also use all available BP readings and treat every clinic BP reading as separate repeated binary assessments.
Change in Home BP | 6 months
  We will also examine change in BP (systolic and diastolic) based on the Home BP measurements from the cellular monitors.
Patient Assessment of Chronic Illness Care (PACIC) | 6 months
  We will collect patient-reported outcomes on a baseline survey at onboarding, with a repeat follow-up survey at 6 months when they exit the study. The Patient Assessment of Care for Chronic Conditions (PACIC) is a 22-item self-measurement of how well patients perceive their chronic condition(s) are being managed by their health care team. Patients fill out a survey of 20 questions regarding elements of the care of their chronic condition(s). Patients answer using a Likert scale of answers ranging from 1-5, with 1 signifying "None of the time" and 5 signifying "Always". The mean is used to find an overall score of the PACIC. The higher scores mean a better outcome.
Krousel-Wood Adherence Scale for medication adherence | 6 months
  We will collect patient-reported outcomes on a baseline survey at onboarding, with a repeat follow-up survey at 6 months when they exit the study. Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4), is a hybrid tool developed to predict pharmacy refill and which captures four domains of adherence behavior: self-efficacy, physical function, intentional medication-taking, and forgetfulness. The 4-item scale categorized participants as low and high adherers using scores at least 1 and less than 1, respectively. The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Lyles, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital/University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No